CLINICAL TRIAL: NCT02221908
Title: ED Decision Making Among Hypotensive Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mespere Lifesciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB1401002513
Record Dates: First submitted 2014-08-18; First posted 2014-08-21 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Hypotension
Keywords: Systolic Blood pressure < 100 mm Hg
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients brought to Hahnemann Hospital ED
  Interventions: Device: Mespere Venus 1000 CVP System

INTERVENTIONS:
Device: Mespere Venus 1000 CVP System

SUMMARY:
The goal of this study is to assess decision making skills of emergency physicians when dealing with hypotensive patients. The hypothesis is that decisions made based on physical exam and vital signs regarding fluid resuscitation by emergency physicians are not statistically equivalent to those that would be made based on the use of a non-invasive CVP measurement

DETAILED DESCRIPTION:
If physicians can make appropriate decisions about the need for fluid resuscitation without CVP measurement, then this skill is worth being passed to physicians in training. Previously it was not possible gather enough information about the response of patients' because of the risk of using indwelling CVP sensors. But now because there is a low risk tool (Venus 1000 System), this study is now practical and safe.

ELIGIBILITY:
Inclusion Criteria:

* All patients >=18 years of age who enter the Emergency Department at Hahnemann Hospital with Systolic Blood pressure < 100 mm Hg

Exclusion Criteria:

* Those patients who are suffering from traumatic injury requiring Level I or Level II trauma evaluations. Example conditions include penetrating injuries to head, torso and proximal extremities.
* Additional exclusion criteria include the presence of an internal jugular or a subclavian central venous line or both external jugular veins being cannulated (attempted or successful) with peripheral IVs.
* Pregnant females will be excluded.
* Subjects under the age of 18 years will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients brough to Hahnemann Hospital ED
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
The correspondence of resuscitation decision and CVP value | At patient admission to ED
  The non-invasive CVP will be measured at the time of initial ordering decision by the ED physician. Afterwards, its relationship to the decision about whether to start intravenous fluid resuscitation will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Handly, MD, Principal Investigator — Drexel University
Locations (1):
- Hahnemann Hospital, Philadelphia, Pennsylvania, United States